CLINICAL TRIAL: NCT04615624
Title: A Randomized Control Trial of Furosemide or Placebo With Usual Antihypertensives in the Antepartum Management of Severe Hypertension With Wide Pulse Pressure
Brief Title: Furosemide vs. Placebo for Severe Antepartum Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Melanie Maykin, MD (Other)
Responsible Party: Sponsor-Investigator, Melanie Maykin, MD, Sponsor-Investigator, Hawaii Pacific Health
Organization: Hawaii Pacific Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-003
Record Dates: First submitted 2020-10-25; First posted 2020-11-04 (Actual); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Pre-Eclampsia; Hypertension in Pregnancy; Pregnancy Complications; Hypertension, Pregnancy-Induced
Keywords: Severe range blood pressure; Pre-eclampsia; Gestational hypertension; Wide pulse pressure; High-risk pregnancy; Pregnancy complications
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Pregnancy Complications | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: After informed consent and upon meeting inclusion criteria, the study personnel will inform pharmacy personnel who will then randomly assigned the patient to groups by opening the next previously prepared sequential and numbered opaque study envelope. The pharmacy staff will send the assigned treatment, which will be administered by the bedside nurse. The vials containing the treatment will be indistinguishable as both furosemide and normal saline placebo are clear, colorless solutions. Thus, the provider, nurse, and patient will be blinded to the treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Furosemide (Experimental): When patient meets inclusion criteria and is randomized to treatment drug, she receives 40mg /4 milliliters (mL) IV furosemide in addition to usual antihypertensive.
  Interventions: Drug: Furosemide
- Placebo (Placebo Comparator): When patient meets inclusion criteria and is randomized to placebo, she receives one dose of 4mL normal saline in addition to usual antihypertensive.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Furosemide — Furosemide, a loop diuretic
  Arms: Furosemide
Other: Placebo — Normal saline
  Arms: Placebo

SUMMARY:
Primary objective: To determine whether the addition of intravenous furosemide with usual antihypertensives is associated with a reduction in mean systolic blood pressure from baseline compared to treatment with placebo plus usual antihypertensives (intravenous labetalol, intravenous hydralazine, or oral immediate release nifedipine) for the management of severe antepartum hypertension.

Secondary objectives:

To determine whether the addition of intravenous furosemide with usual antihypertensives is associated with a reduction in mean diastolic blood pressure compared to treatment with placebo plus usual antihypertensives listed above.

DETAILED DESCRIPTION:
Blood pressure is a measure of blood flow and resistance in blood vessels. In normal pregnancy, total blood volume increases while systemic vascular resistance decreases, thereby leading to an overall reduction in blood pressure with return to baseline at term. Hypertensive disorders in pregnancy, including preeclampsia, are a polymorphic syndrome characterized by elevated blood pressures which can affect multiple organ systems. Although the exact mechanism of preeclampsia has yet to be determined, previous studies have shown that there may be two distinct phenotypes - one characterized by vasoconstriction and diminished micro-circulation and the other involving a hyperdynamic high cardiac output state.

Given its potential for both significant maternal and fetal morbidity, hypertensive disorders in pregnancy comprise a substantial proportion of antepartum admissions. Management of acute severe hypertension (systolic blood pressure greater than or equal to 160 or diastolic blood pressure greater than or equal to 110) is important to reduce the risk of stroke, hypertensive encephalopathy, placental abruption, and heart failure or myocardial infarction. In the antepartum and intrapartum period, the use of antihypertensives including labetalol, nifedipine, and hydralazine have been well-described. Despite these options for blood pressure control, preeclampsia can be a progressive disorder that may not respond to the aforementioned agents.

In preeclampsia manifested by high blood volume due to salt and water retention rather than vasoconstriction, standard antihypertensives may be less effective. Furosemide is a commonly used diuretic that can lower blood pressure by inhibiting the absorption of sodium, chloride, and water, thereby decreasing the volume of blood that the heart pumps. The onset of action of action of IV furosemide is 5 minutes, with peak effect at 30 minutes, and duration of action of 2 hours.

Previous studies have demonstrated the safety and efficacy of furosemide to treat preeclampsia in the antepartum and postpartum period as well as its utility in treating heart failure in pregnant women. To our knowledge, no randomized studies exist that investigate the use of furosemide in treating hypertension in the antepartum period. We aim to determine the utility of the addition of furosemide to usual antihypertensives in this clinical setting.

This will be a prospective double-blinded randomized placebo control trial of women with a diagnosis of preeclampsia with severe features at ≥20 weeks of gestation with persistent antepartum hypertension (sustained systolic blood pressure ≥160 or diastolic blood pressure ≥110 mmHg) and a wide pulse pressure (>60 mmHg) who meet all inclusion criteria and have no exclusion criteria. It is routine that laboratory studies are performed on admission for all women with hypertensive disorders. If electrolyte disturbances exist, therapy will not be initiated unless the electrolyte is normalized or repleted.

After informed consent and upon meeting inclusion criteria with severe range hypertension with wide pulse pressure, the study personnel will inform pharmacy personnel who will then randomly assigned the patient to groups by opening the next previously prepared sequential and numbered opaque study envelope. Participants will be randomized to furosemide plus an antihypertensive versus placebo containing normal saline and an antihypertensive. The pharmacy staff will send the assigned treatment, which will be administered by the bedside nurse. The vials containing the treatment will be indistinguishable as both furosemide and normal saline placebo are clear, colorless solutions. Thus, the provider, nurse, and patient will be blinded to the treatment. The choice of antihypertensive will be determined by the primary obstetric provider. At our institution, this will be one or more of the recommended medications for urgent blood pressure control as outlined by the American College of Obstetricians and Gynecologists Practice Bulletin on gestational hypertension and preeclampsia. These include IV labetalol, IV hydralazine, or immediate-release oral nifedipine. As meta-analyses have not shown that one of the aforementioned antihypertensives is superior than another, and all are reasonable options, the choice of antihypertensive will be left up to the obstetric provider. This will also improve the generalizability of the study as it does not interfere with what is typically done in clinical practice.

As a procedure of the study, patients will have their blood pressure recorded at least every 15 minutes up to one hour after administration of the study drug. Thereafter, as part of routine care, patients in both groups will receive similar antepartum surveillance, including blood pressure and pulse assessment every four hours or more frequently if vital signs are abnormal, daily weight measurement, and daily urinary output measurements.

Study Procedures

1. Antepartum patient diagnosed with a hypertensive disorder in pregnancy.
2. Patient approached for study participation and informed consent obtained if interested.
3. Patient develops severe range BP (systolic blood pressure > or = 160 and/or diastolic blood pressure> or =10) with increased pulse pressure (>60mmHg). This will be considered baseline BP.
4. When ordering provider's choice of antihypertensive, pharmacy notified that patient is study participant and randomizes patient by choosing from sequential opaque envelope.
5. a. Patient randomized to treatment arm and receives 40mg /4 milliliters IV furosemide in addition to usual antihypertensive.

   b. Patient randomized to placebo and receives 4 milliliters normal saline in addition to usual antihypertensive.
6. Blood pressure check every 15 minutes after administration of furosemide/placebo for four recordings (15, 30, 45, 60 minutes)

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older
* Subjects with intrauterine pregnancy at or beyond 20 weeks of gestation
* Subjects with a diagnosis of hypertensive disorder in pregnancy
* Subjects with persistent (on repeat BP check 15 min apart) severe range blood pressure recordings (systolic BP greater than or equal to 160 or diastolic greater than or equal to BP 110) with wide pulse pressure (>60 mmHg)
* Subject able to provide informed consent

Exclusion Criteria:

* Subjects less than 18 years of age
* Subjects with intrauterine pregnancy less than 20 weeks of gestation
* Subjects with known fetal anomaly
* Subjects with hypokalemia (K <3.0 milliequivalent per liter) on admission
* Subjects with anuria (<50 milliliters urine in 24 hours) or renal failure
* Subjects previously taking diuretics or potassium supplements for any reason
* Subjects with a known allergy/adverse reaction to furosemide
* Subjects who are unable to understand and/or sign the informed consent
* Subjects who are in active labor defined as 6 centimeters of cervical dilation or more
* Subjects who have an epidural (neuraxial anesthesia) in place

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Tsai, MD, Principal Investigator — Maternal-Fetal Medicine Faculty
Locations (1):
- Kapiolani Medical Center for Women and Children, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: Yes
Will individual participant data be available (including data dictionaries)? Individual participant data will be made available.
  What data in particular will be shared? Individual participant data that underlie the results reported any future manuscript, after deidentification (text, tables, figures, and appendices).
  What other documents will be available? There are no plans for additional documents to be made available.
  When will data be available (start and end dates)? Beginning 9 months and ending 36 months following any publication.
  With whom? Researchers who provide a methodologically sound proposal.
  For what types of analyses? To achieve aims in the approved proposal.
Time Frame: Beginning 9 months and ending 36 months following any publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Grindheim G, Estensen ME, Langesaeter E, Rosseland LA, Toska K. Changes in blood pressure during healthy pregnancy: a longitudinal cohort study. J Hypertens. 2012 Feb;30(2):342-50. doi: 10.1097/HJH.0b013e32834f0b1c. PMID 22179091
- [Background] Phillips JK, Janowiak M, Badger GJ, Bernstein IM. Evidence for distinct preterm and term phenotypes of preeclampsia. J Matern Fetal Neonatal Med. 2010 Jul;23(7):622-6. doi: 10.3109/14767050903258746. PMID 20482241
- [Background] Easterling TR, Benedetti TJ, Schmucker BC, Millard SP. Maternal hemodynamics in normal and preeclamptic pregnancies: a longitudinal study. Obstet Gynecol. 1990 Dec;76(6):1061-9. PMID 2234714
- [Background] ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003018. PMID 30575675
- [Background] https://www.uptodate.com/contents/furosemide-drug information?search=furosemide&source=panel_search_result&selectedTitle=1~148&usage_type=panel&kp_tab=drug_general&display_rank=1
- [Background] Tamas P, Hantosi E, Farkas B, Ifi Z, Betlehem J, Bodis J. Preliminary study of the effects of furosemide on blood pressure during late-onset pre-eclampsia in patients with high cardiac output. Int J Gynaecol Obstet. 2017 Jan;136(1):87-90. doi: 10.1002/ijgo.12019. Epub 2016 Nov 3. PMID 28099709
- [Background] Ascarelli MH, Johnson V, McCreary H, Cushman J, May WL, Martin JN Jr. Postpartum preeclampsia management with furosemide: a randomized clinical trial. Obstet Gynecol. 2005 Jan;105(1):29-33. doi: 10.1097/01.AOG.0000148270.53433.66. PMID 15625138
- [Background] Duley L, Meher S, Jones L. Drugs for treatment of very high blood pressure during pregnancy. Cochrane Database Syst Rev. 2013 Jul 31;2013(7):CD001449. doi: 10.1002/14651858.CD001449.pub3. PMID 23900968
- [Background] Committee on Obstetric Practice. Committee Opinion No. 692: Emergent Therapy for Acute-Onset, Severe Hypertension During Pregnancy and the Postpartum Period. Obstet Gynecol. 2017 Apr;129(4):e90-e95. doi: 10.1097/AOG.0000000000002019. PMID 28333820
- [Derived] Maykin MM, Mercer E, Saiki KM, Kaneshiro B, Miller CB, Tsai PS. Furosemide to lower antenatal severe hypertension: a randomized placebo-controlled trial. Am J Obstet Gynecol MFM. 2024 Apr;6(4):101348. doi: 10.1016/j.ajogmf.2024.101348. Epub 2024 Mar 12. PMID 38485054

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Furosemide | Placebo
Started | 33 | 32
Completed | 33 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Furosemide | Placebo | Total
Number analyzed (Participants) | 33 | 32 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 32 | 65
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 33 | 32 | 65
  Sex: Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 7 | 6 | 13
  Race/Ethnicity: Filipino | 16 | 12 | 28
  Race/Ethnicity: Native Hawaiian | 3 | 4 | 7
  Race/Ethnicity: Micronesian | 1 | 4 | 5
  Race/Ethnicity: White | 5 | 1 | 6
  Race/Ethnicity: All others | 1 | 5 | 6
obese [Count of Participants; unit: Participants] | 14 | 18 | 32
insurance [Count of Participants; unit: Participants]
  Commercial | 24 | 18 | 42
  Public | 9 | 14 | 23
nulliparous [Count of Participants; unit: Participants] | 18 | 14 | 32
twin pregnancy [Count of Participants; unit: Participants] | 2 | 2 | 4
hypertension subtype [Count of Participants; unit: Participants]
  new-onset | 14 | 18 | 32
  pre-existing | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Mean Systolic Blood Pressure During Hour After Study Drug
Description: Mean systolic blood pressure during hour after study drug administration.
Time Frame: 0 minutes to 60 minutes post-dose
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
mmHg | 147 (14.8) | 152 (13.8)

2. Secondary Outcome: Mean Diastolic Blood Pressure During Hour After Study Drug
Description: Mean diastolic blood pressure during the 1-hour period after drug administration.
Time Frame: 0 minutes to 60 minutes post-dose
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
mmHg | 88 (10.8) | 87 (9.3)

3. Secondary Outcome: Change From Qualifying Systolic Blood Pressure
Description: Change from qualifying systolic blood pressure (qualifying SBP-mean SBP during hour after intervention) where qualifying systolic blood pressure refers to a severe range SBP (>=160 millimeters of mercury (mmHg)) for at least 15 minutes.
Time Frame: 0 minutes to 1 hour post-dose
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
mmHg | -26 (13.9) | -24 (15.5)

4. Secondary Outcome: Change From Qualifying Diastolic Blood Pressure
Description: Change from qualifying diastolic blood pressure (qualifying DBP-mean DBP during hour after intervention) where qualifying diastolic blood pressure refers to a severe range DBP (>=110 millimeters of mercury (mmHg)) for at least 15 minutes.
Time Frame: 0 minutes to 1 hour post-dose
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
mmHg | -12 (7.6) | -11 (8.9)

5. Secondary Outcome: Pulse Pressure at 2 Hours After Study Drug.
Description: Pulse pressure at 2 hours after study drug.
Time Frame: 2 hours post-dose
Population: Not every participant had their blood pressure and thus pulse pressure checked at 2 hours which is a limitation of the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 27 | 22
mmHg | 55 (12.5) | 67 (15.1)

6. Secondary Outcome: Systolic Blood Pressure at 2 Hours After Study Drug
Description: Systolic blood pressure at 2 hours after study drug
Time Frame: 2 hours post-dose
Population: Not every participant had their blood pressure checked at 2 hours which is a limitation of the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 27 | 22
mmHg | 139 (18.5) | 154 (18.4)

7. Secondary Outcome: Diastolic Blood Pressure at 2 Hours After Study Drug
Description: Diastolic blood pressure at 2 hours after study drug
Time Frame: 2 hours post-dose
Population: Not every participant had their blood pressure checked at 2 hours which is a limitation of the study.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 27 | 22
mmHg | 84 (12.5) | 87 (10.5)

8. Other Pre Specified Outcome: Gestational Age at Delivery
Description: Gestational age in weeks and days at the time of birth
Time Frame: at the time of birth
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
weeks | 34.1 (2.9) | 34 (3.1)

9. Other Pre Specified Outcome: Time From Admission to Delivery
Description: Time in days and hours from admission to birth
Time Frame: at the time of delivery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
days | 2.3 [1.1 to 14.6] | 3.7 [1.1 to 11.2]

10. Other Pre Specified Outcome: Time From Treatment to Delivery
Description: Time in days and hours from treatment to birth
Time Frame: at the time of delivery
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
days | 2.1 [.8 to 10.9] | 1.8 [.7 to 6.5]

11. Other Pre Specified Outcome: Induction of Labor
Description: Number of women who required induction of labor
Time Frame: at the time of induction of labor
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
Participants | 7 | 4

12. Other Pre Specified Outcome: Mode of Delivery
Description: Type of delivery
Time Frame: at time of delivery
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
Participants
  spontaneous vaginal delivery | 9 | 8
  operative vaginal delivery | 0 | 2
  Cesarean section | 24 | 22

13. Other Pre Specified Outcome: Eclampsia
Description: Number of women who developed seizure
Time Frame: at time of hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
Participants | 0 | 0

14. Other Pre Specified Outcome: Low Apgar Scores of Neonate (Apgar Score <7 at 5 Min)
Description: Neonatal clinical assessment (Apgar is not an abbreviated term). Minimum value 0; maximum value 9; Tool is used for assessment and not an accurate prognostic tool to predict outcomes.
Time Frame: at 5 minutes after delivery
Measure: Number; unit: neonates
Units Other Than Participants: neonates
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
Number analyzed (neonates) | 35 | 34
neonates | 3 | 3

15. Other Pre Specified Outcome: Newborns Admitted to Intensive Care Nursery
Description: Neonatal Intensive Care Unit admission
Time Frame: assessed from time of delivery until discharge since neonates can be admitted to the NICU at any time during this interval if issues arise.
Measure: Number; unit: neonates
Units Other Than Participants: neonates
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
Number analyzed (neonates) | 35 | 34
neonates | 24 | 25

16. Other Pre Specified Outcome: Time to Achieve First Non-severe BP (m)
Description: Time to achieve first non-severe BP (m)
Time Frame: Assessed from time of severe range blood pressure to time at resolution of severe range blood pressure. Reported at time of resolution of severe range blood pressure.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
minutes | 44 [23 to 75] | 46 [30 to 76]

17. Other Pre Specified Outcome: Number of Participants Who Required Additional Antihypertensive Agents in an Hour After Allocation
Description: Were any additional antihypertensive agents in hour after allocation
Time Frame: Assessed from 0 minutes to 1 hour post-dose, 1-hour post-dose reported
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
Participants | 9 | 7

18. Other Pre Specified Outcome: Latency Until Next First-line Antepartum Antihypertensive Agents
Description: time until next first-line antepartum antihypertensive agent given
Time Frame: 0 minutes to delivery of baby (72 hours post-dose)
Population: Those who required additional medication (not all participants required additional antihypertensive medication).
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 23 | 22
hours | 10.8 [.8 to 31.1] | 3.2 [.4 to 25.9]

19. Other Pre Specified Outcome: Discharged Without Delivery
Description: proportion of participants who were discharged prior to delivery of the baby
Time Frame: at time of hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
Participants | 6 | 3

20. Other Pre Specified Outcome: Length of Stay
Description: length of stay
Time Frame: at time of hospital discharge
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
days | 6.1 [4.3 to 12.5] | 7.3 [4.1 to 7.3]

21. Other Pre Specified Outcome: Birthweight
Description: weight of baby at birth
Time Frame: at time of birth
Measure: Mean (Standard Deviation); unit: grams
Units Other Than Participants: neonates
Arm/Group | Furosemide | Placebo
Number analyzed (Participants) | 33 | 32
Number analyzed (neonates) | 35 | 34
grams | 1921 (534.7) | 2070 (796.4)

ADVERSE EVENTS:
Time Frame: 1 year and 3 months
Description: Adverse events include allergic reaction to the intervention, hypotension, illness thought to be caused by the intervention, and death.
Arm/Group | Furosemide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 0/33 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/24/NCT04615624/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT04615624/ICF_001.pdf